CLINICAL TRIAL: NCT06312839
Title: Preoperative Arterial Embolization Before Oncologic Esophagectomy as a Technique for Ischemic Gastric Conditioning : a Retrospective Monocentric Comparative Study
Brief Title: Preoperative Arterial Embolization Before Oncologic Esophagectomy as a Technique for Ischemic Gastric Conditioning
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN032024/CHUSTE
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer
Keywords: Embolization; Ischemic conditioning; Esophagectomy; Lewis Santy; Anastomotic leakage
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Esophagectomy alone
  Interventions: Other: Collecting data from the medical record
- Study Group: Preoperative ischemic conditioning before esophagectomy
  Interventions: Other: Collecting data from the medical record

INTERVENTIONS:
Other: Collecting data from the medical record — Collecting data from the medical record:
  * Gastroepiploic artery diameter before and after ischaemic preconditioning
  * Postoperative mortality
  * Complications related to embolisation and surgery
  * Length of stay in intensive care unit and total length of hospital stay

SUMMARY:
This retrospective monocentric comparative study aims to assess the efficacy of preoperative ischemic conditioning, in preventing anastomotic leakage in esophageal cancer surgery. Two groups were included : a surgery-alone group (control group) and a PreopAE group (study group) treated with an embolization procedure before esophagectomy. Collected data included patient characteristics, embolization procedure details, surgical outcomes, and postoperative complications.

The primary outcome was the efficacy of preoperative ischemic conditioning in preventing anastomotic leakage, assessed through CT scans. Secondary outcomes included analyzing safety of ischemic gastric conditioning, hypertrophy of the gastroepiploic artery in embolized patients and comparing hospital stay length and postoperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years with an indication for surgical esophagectomy with cervical anastomosis using the Lewis Santy technique or three stages approach.

Exclusion Criteria:

* Esophagectomy for ischemic or caustic oesophagitis, and patients lost for follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic oesophageal cancer, eligible for curative surgery by oesophagectomy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of the effectiveness of preoperative ischaemic conditioning in reducing anastomotic leakage in patients undergoing oesophagectomy. | Day : 90
  Radiological confirmation by thoracoabdominal CT scan with oral contrast showing dehiscence of the oesophagastric anastomosis will be sought.

SECONDARY OUTCOMES:
Measurement of the effectiveness of preoperative ischaemic conditioning in reducing anastomotic leakage in patients undergoing oesophagectomy. | Day : 90
  Dehiscence confirmed by the surgeon during a repeat operation will be sought.
Measurement of the effectiveness of preoperative ischaemic conditioning in reducing anastomotic leakage in patients undergoing oesophagectomy. | Day : 90
  Endoscopic confirmation of an anastomotic leak will be sought.
Safety of ischemic gastric conditioning | Day : 90
  Safety of ischaemic gastric filling will be analysed on the basis of imaging and data recordings.
Hypertrophy of the gastroepiploic artery | Day : 90
  Hypertrophy of the gastroepiploic artery in embolized patients will be analysed on the basis of imaging and data recordings.
Comparing hospital stay length | Day : 90
  Hospital stay length will be analysed on the basis of data recordings.
Comparing postoperative mortality | Day : 90
  Postoperative mortality will be analysed on the basis of data recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi GRANGE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No